CLINICAL TRIAL: NCT05153603
Title: Outcomes of First-line Olaparib Mono-maintenance Therapy in Newly Diagnosed Ovarian Cancer Patients With tBRCA Wild-type Tumors: a Realworld Study
Brief Title: Outcomes of First-line Olaparib Mono-maintenance therapy-a Multicenter, Retrospective Study Using Data From Real-world Clinical Setting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-20-20889-02
Record Dates: First submitted 2021-12-08; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Neoplasms
Keywords: tBRCA， olaparib
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Olaparib mono-maintenance therapy group: Olaparib monotherapy in clinical practice and will be conducted in patients with tBRCAwt newly diagnosed high grade epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy following the standard of care from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required) at tertiary-referral university hospitals and main cancer centers in China.
  Interventions: Drug: Olaparib mono-maintenance therapy

INTERVENTIONS:
Drug: Olaparib mono-maintenance therapy — Olaparib mono-maintenance therapy in patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III-IV) ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer is defined as drug exposure. At least one dose of olaparib tablets monotherapy as maintenance therapy will be required.

SUMMARY:
Four phase III trials in ovarian cancer consistently showed that front-line poly(ADP-ribose) polymerase (PARP) inhibition can significantly improve progression-free survival. Based on these findings, current clinical guidelines recommend the olaparib + bevacizumab combination as a maintenance therapy for ovarian cancer patients with BRCA1/2 wild-type or unknown mutation status who have a complete response (CR)/ partial response (PR) after completing bevacizumab-containing first-line therapy. However, bevacizumab is not a NATIONAL MEDICAL PRODUCTS ADMINSTRATION（NMPA）-approved agent for ovarian cancer patients. In this setting, olaparib mono-maintenance therapy has been implemented among patients with BRCA-wild type tumors in clinical practice in China.

DETAILED DESCRIPTION:
The main objective is to evaluate the outcome of olaparib-based maintenance therapy by proportion of patients alive and progression free at 1 year (1-yr PFS rate) We hypothesize that olaparib monotherapy could be beneficial for tBRCAwt high-grade serous ovarian cancer (HGSOC) patients who are treated with platinum-based first-line chemotherapy.

The secondary objectives are to evaluate the outcomes of olaparib-based maintenance therapy by: 1) 2-yr PFS rate; 2) median PFS; 3) median Time to First Subsequent Therapy or death (mTFST) ; 4) post-progression treatment after first progression; 5) reason for olaparib dose adjustment, dose interruptions, and dose discontinuations; 6) Reason for use of concomitant therapy.

The exploratory objective is to evaluate the status quo of genetic testing, R0 resection and related outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they met all the following criteria:

* Female Patients must be ≥18 years old at diagnosis.
* Patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III-IV) ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer and received olaparib from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required).
* Patients must have a tumor BRCA testing result which is tBRCAwt, defined as tumor BRCA wild type (patients without evidence of BRCA 1 and/or BRCA 2 deleterious or suspected deleterious mutations).
* Patients who have completed first-line platinum-based chemotherapy and were in clinical complete response (CR) or in partial response (PR).
* Patients who were still in CR or PR before receiving maintenance therapy.
* Patients who received at least one dose of olaparib tablets monotherapy as maintenance therapy within three months after platinum-based chemotherapy and without disease progression.

Exclusion Criteria:

Patients are excluded if any of the following factors were present:

* Patient with multiple primary cancers as reported in EMR.
* Concomitant any anti- cancer therapy (chemotherapy, immunotherapy, hormonal therapy (Hormone replacement therapy (HRT) is acceptable), radiotherapy, biological therapy or other novel agent) during Olaparib maintenance.
* Any previous treatment with PARP inhibitor.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases.
* Any other concerns related to decreased efficacy and safety of maintenance therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HGSOC who started first-line PARPi maintenance therapy from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required) will be identified from the electronic medical record system.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
1-yr PFS rate | 12 months after date of first dose
  The main objective is to evaluate the outcome of olaparib-based maintenance therapy by proportion of patients alive and progression free at 1 year.

SECONDARY OUTCOMES:
2-yr PFS rate | 24 months after date of first dose
  The proportion of patients alive and progression free by 2 years by investigator assessed clinical progression
Median PFS | Median time from date of first dose until disease progression
  Median time from date of first dose until disease progression per clinical progression (mPFS) as assessed by the investigator at local site or death due to any cause (if this occurs before disease progression)
mTFST | Median time from date of first dose to the earlier of start date of the first subsequent anti-cancer therapy after discontinuation of treatment or death due to any cause
  Median Time to First Subsequent Therapy or death
post-progression treatment after first progression | The proportion of patients receiving each treatment after first progression
  The proportion of patients receiving each treatment after first progression
Reason for olaparib dose adjustment, dose interruptions, and dose discontinuations | The proportion of olaparib dose adjustment, dose interruptions, and dose discontinuations
  The proportion of olaparib dose adjustment, dose interruptions, and dose discontinuations
Reason for use of concomitant therapy | The proportion of concomitant therapy
  The proportion of concomitant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-qiu Lin, MD, PhD,Professor, Study Chair — Department of Gynecologic Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-sen University; Jing Li, MD, PhD,Professor, Principal Investigator — Department of Gynecologic Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-sen University